CLINICAL TRIAL: NCT05813197
Title: Leaving Care - a Comparison Study of Implementation, Change Mechanisms, and Effects of Transition Services for Youth Leaving Out-of-home Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jonkoping University (Other)
Collaborators: Lund University (Other); Göteborg University (Other)
Responsible Party: Principal Investigator, Tina M. Olsson, Associate Professor, Jonkoping University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-01352
Record Dates: First submitted 2023-03-21; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Self Efficacy; Mental Health Wellness 1; Help-Seeking Behavior; Frustration; Satisfaction; Health Behavior
MeSH Terms: conditions — Help-Seeking Behavior; Personal Satisfaction; Health Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group will receive the test intervention My Choice-My Way!
  Interventions: Behavioral: My Choice - My Way!
- Control (Active Comparator): This group will receive usual services
  Interventions: Behavioral: Usual services

INTERVENTIONS:
Behavioral: My Choice - My Way! — Support intervention for adolescents (15+) in out-of-home care (foster care, group home care, supported living, institutional care, etc). 16-19 sessions with a MCMW coach, 4-8 months, weekly to bi-weekly sessions.
  Arms: Intervention
Behavioral: Usual services — Usual services
  Arms: Control

SUMMARY:
The purpose of this project is to increase understanding of the development, implementation and effectiveness of interventions for young people transitioning from societal care to independent living. The project examines the effect of interventions and how change mechanisms relate to a range of outcomes.

DETAILED DESCRIPTION:
The purpose of this project is to increase the empirical understanding of the development, implementation and effectiveness of interventions for young people transitioning from societal care to independent living. The project examines the effect of interventions and how change mechanisms relate to a range of outcomes. In a pilot project, the investigators developed an intervention in collaboration with municipal social workers, section heads and organizational developers. In another pilot project, the investigators studied whether the content of empirically tested interventions in the USA can be generalized to a Swedish context. These two projects have resulted in a Swedish intervention: My choice - my way! Previous research shows that young people who are placed in social care are a particularly vulnerable group. Swedish social places little attention to what happens to prepare young people for leaving care. There are currently no interventions in Sweden that have empirical support of their effectiveness for this group. The aim of the project is to develop practical and empirical understanding of how interventions for young people placed in societal care in Sweden can be developed and implemented. The project takes place in close collaboration with municipalities and other youth serving organizations. Short-term, long-term and implementation effects are investigated by comparing My choice - my way! with usual services. The comparisons will shed light on practice components and change mechanisms related to outcomes and thus important to take into account in the future development of interventions. The outcomes will shed light on a range of self-reported outcomes, as well as register-based outcomes such as education, employment and crime. The analyses also include health economic outcomes. In addition, the attitudes of social workers and youth and organizational implementation initiatives will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Living in out-of-home care
* 15 years or older

Exclusion Criteria:

* none

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-10-02 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Needs Satisfaction and Frustration Scale (NSFS) | 8 months
  Autonomy, relatedness, competence
General Self-Efficacy Scale (GSE-10) | 8 months
  Self-efficacy
Resilience Scale (RS-14) | 8 months
  Resilience
Needs Satisfaction and Frustration Scale (NSFS) | 17 months
  Autonomy, relatedness, competence
General Self-Efficacy Scale (GSE-10) | 17 months
  Self-efficacy
Resilience Scale (RS-14) | 17 months
  Resilience

SECONDARY OUTCOMES:
General Health Questionnaire (GHQ-12) | 8 months
  Measure of psychological distress
General Help-Seeking Questionnaire (GHSQ) | 8 months
  Intentions, quantity, and quality of help seeking
Social Support Questionnaire (SSQ-6) | 8 months
  Social Support
Daily Routines (DR-18) | 8 months
  Daily Routine
General Health Questionnaire (GHQ-12) | 17 months
  Measure of psychological distress
General Help-Seeking Questionnaire (GHSQ) | 17 months
  Intentions, quantity, and quality of help seeking
Social Support Questionnaire (SSQ-6) | 17 months
  Social Support
Daily Routines (DR-18) | 17 months
  Daily Routine

OTHER OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8, T2) | 8 months
  General satisfaction with services

CONTACTS AND LOCATIONS:
Overall Officials: Tina M Olsson, PhD, Principal Investigator — Jonkoping University
Locations (1):
- Jönköping University, Jönköping, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
no plan as of yet

REFERENCES:
- [Derived] Skoog T, Bergstrom M, Karlsson M, Olsson TM. Study protocol for leaving care-A comparison study of implementation, change mechanisms and effectiveness of transition services for youth. PLoS One. 2024 Feb 8;19(2):e0293952. doi: 10.1371/journal.pone.0293952. eCollection 2024. PMID 38329996